CLINICAL TRIAL: NCT02185144
Title: The PFT Intervention: Linking Triply Diagnosed Inpatients to Community Care
Brief Title: PATH For Triples Study: Medication and Lifestyle Adherence for HIV+ Patients
Acronym: PFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01DA036503-01A1 (NIH)
Record Dates: First submitted 2014-06-30; First posted 2014-07-09 (Estimated); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: HIV
Keywords: HIV, mental health, substance abuse
MeSH Terms: conditions — Psychological Well-Being; Substance-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PATH for Triples (PFT) (Experimental): The Nurse Health Navigator (NHN) meets at least weekly with the experimental participants to implement the adherence component of PFT using approaches tailored to the communication and comprehension of the person that includes memory aids, education regarding side effects and other treatment aspects, engagement with participants' social networks and treatment providers, and active community outreach. PFT will be implemented for 6 months and participants will be followed for an additional 3 months to allow examination of potential decay of the intervention after it is withdrawn.
  Interventions: Behavioral: PATH For Triples
- Treatment as Usual (TAU) (Placebo Comparator): Participants in the the Treatment as Usual (TAU) group receive usual treatment after inpatient care.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: PATH For Triples — In addition to providing weekly home-health nursing focused psycho-education aimed at insuring adherence to drug treatment regimen, the nurse health navigator model provided in PFT combines continuous and integrated care across mental health, substance abuse, and infectious disease provides. The nurses will accompany the patient to appointments, or make collateral contacts with other care providers. Often the nurses serve as intermediaries and ensure accurate and timely information exchange. Their specialized training also allows them to monitor side effects of medications and advocate for the patients with their various specialty providers. A treatment cascade approach is utilized when the patient is non-adherent to treatment allowing for increased patient monitoring.
  Arms: PATH for Triples (PFT)
Behavioral: Treatment as Usual — Control subjects receive enhanced TAU care which will consist of the opportunity to complete the full complement of baseline instruments that will then be shared with their outpatient mental health case manager to facilitate linkage with needed MH, SA, and ID care
  Arms: Treatment as Usual (TAU)

SUMMARY:
The PATH for Triples (PFT) Study is an effectiveness trial comparing a nurse health navigator (NHN) model for HIV+ persons with severe mental illness and substance abuse (i.e., triply diagnosed) with Treatment as Usual (TAU). The team completed a Phase II trial of the nurse health navigator model for HIV+ persons with severe mental illness that showed the intervention was effective. The investigators are now testing the intervention in a real world setting with patients recruited from psychiatric and substance abuse inpatient units in Philadelphia using a longitudinal design. The intervention is set up as a cascade where non-adherent patients receive additional visits from the study nurses. It is hypothesized that patients assigned to the NHN will have better medication compliance, reduced viral loads and improved CD4 counts compared to patients assigned to TAU. It is also hypothesized that the PFT intervention group will be more cost effective compared to TAU. This group of triply diagnosed patients are at very high risk of negative health outcomes and secondary transmission of HIV and, therefore, the study is of high public health significance.

DETAILED DESCRIPTION:
In response to PA-12-281, HIV/AIDS, Drug Use, and Vulnerable Populations in the US (R01), we are conducting an effectiveness trial among persons triply diagnosed (mental illness, substance abuse, HIV) recruited from inpatient psychiatric units in Philadelphia. Despite general recognition that persons with serious mental illness (SMI) are at heightened risk to contract and transmit human immunodeficiency virus (HIV), systematic HIV testing in mental health settings is rare. Using discarded blood samples over a six-month period, our research team found in excess of 10% HIV seroprevalence in two inpatient psychiatric units in Philadelphia. We argued then that HIV testing should be routinely conducted in those settings. In a five-year longitudinal effectiveness trial, we will identify HIV positive SMI inpatients through rapid testing. Those who are newly diagnosed or who were previously diagnosed but not currently engaged in HIV treatment and who also are substance using will be offered an opportunity to participate in a randomized community trial. Previously, we have conducted a Phase II trial of PATH for Positives (PFP) in which we observed broad and far-reaching effects of an intervention utilizing a nurse health navigator (NHN) model for HIV+ SMI clients. The current study builds on what we learned previously to provide a nurse health navigator (NHN) model as integrated treatment of the targeted individuals in "real world" conditions and to monitor the implementation of PATH for Triples (PFT). The target population is arguably among the highest risk patient populations for poor treatment outcomes. Based on past experience, we expect to enroll about 75% of those eligible on a rolling basis, or ~240 participants who will then be randomized. This will yield ~120 PFT and ~120 Treatment as Usual (TAU) participants over a 36-month recruitment window before attrition. A similar population in PFP resulted in a 17% attrition rate, so we estimate complete data for at least 75% of participants resulting in a complete dataset of ~180 participants (90 PFT, and 90 TAU). PFT participants will receive NHN services for 6 months. Data will be collected at baseline, 3, 6, and 9 months for each participant. Participants will be followed longitudinally for an additional 3 months post intervention to measure any decay of the intervention after it is withdrawn. Experimental participants will begin PFT while still receiving inpatient services and the project nurses will participate in discharge planning and facilitate linkage to Mental Health (MH), Substance Abuse (SA), and Infectious Disease (ID) care in the Philadelphia community. The NHN will also meet at least weekly with the experimental participants to implement the adherence component of PFT using approaches tailored to the communication and comprehension of the person that includes memory aids, education regarding side effects and other treatment aspects, engagement with participants' social networks and treatment providers, and active community outreach. We expect better retention in treatment for PFT participants and improvement in other outcomes including viral load, CD4, indicators of psychological and social functioning, and cost effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* 18 or older;
* HIV+;
* Newly diagnosed w/HIV or not currently in care for HIV;
* Receiving psychiatric inpatient care;
* Have a serious mental illness;
* Have co-occurring substance use or abuse;
* Ability to speak English;
* Ability to provide informed consent;
* Willingness to provide locator information;
* Willingness to be randomized to PFT or TAU.
* Resident of the City of Philadelphia

Exclusion Criteria:

* HIV-;
* Persons who are unable to provide informed consent;
* Inability to speak English;
* Not willing to provide locator information;
* Not competent to provide informed consent;
* If HIV status is unknown, they refused to be tested;
* Not a resident of the City of Philadelphia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2014-02; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Change in HIV status based on viral load from baseline through 9 months | Baseline, 3, 6, 9 months
  Change in viral load based on collection of blood specimens at baseline, 3, 6 and 9 months
Change in HIV status based on CD4 count from baseline through 9 months | Baseline, 3, 6, 9 months
  Change in CD4 count based on collection of blood specimens at baseline, 3, 6 and 9 months

SECONDARY OUTCOMES:
Medical, psychiatric and substance abuse services used by study participants over the 9-month duration of the study using Medicaid Claims Data | 9 months
  To assess the cost effectiveness of PFT compared to Treatment as Usual using Medicaid Claims Data.
Change in HIV knowledge and intentions from baseline through 9 months using the HIV Intention and Knowledge Measure | Baseline, 3, 6, 9 months
Change in HIV risk behaviors based on the Risk Assessment Battery from baseline through 9 months | Baseline, 3, 6, 9 months
Change in mental health functioning using the BASIS24 from baseline through 9 months | Baseline, 3, 6, 9 months
Change in alcohol use using the ASSIST Measure from baseline through 9 months | Baseline, 3, 6, 9 months
Change in alcohol use based on the Seek, Test, Treat and Retain for Vulnerable Populations: Data Harmonization Measure from baseline through 9 months | Baseline, 3, 6, 9 months
Change in drug use based on the ASSIST from baseline through 9 months | Baseline, 3, 6, 9 months
Change in drug use based on the Seek, Test, Treat and Retain for Vulnerable Populations: Data Harmonization Measure from baseline through 9 months | Baseline, 3, 6 and 9 months
Change in quality of life based on the SF12 from baseline through 9 months | Baseline, 3, 6 and 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Blank, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Blank MB, Himelhoch SS, Balaji AB, Metzger DS, Dixon LB, Rose CE, Oraka E, Davis-Vogel A, Thompson WW, Heffelfinger JD. A multisite study of the prevalence of HIV with rapid testing in mental health settings. Am J Public Health. 2014 Dec;104(12):2377-84. doi: 10.2105/AJPH.2013.301633. Epub 2014 Feb 13. PMID 24524493